CLINICAL TRIAL: NCT01148459
Title: Safety and Immunogenicity Study of GSK Biologicals' Plasmodium Falciparum Malaria Vaccine 257049 Administered to HIV Infected Infants and Children
Brief Title: Safety and Immunogenicity of GSK Biologicals' Investigational Malaria Vaccine in HIV Infected Infants and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 112745
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2017-05

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; schedule; HIV; malaria vaccine; EPI; Africa
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Rabies Vaccines; lactitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group A (Experimental): Infants enrolled to this group will receive 3 doses of the experimental vaccine.
  Interventions: Biological: GSK Biological's Investigational Malaria Vaccine 257049
- Group B (Active Comparator): Infants enrolled to this group will receive 3 doses of the rabies comparator vaccine.
  Interventions: Biological: Human Diploid Cell Vaccine (HDCV) or Purified Vero Cell Rabies Vaccine (PVRV, Verorab) (Aventis Pasteur);; Biological: Purified Chick Embryo Cell Culture (PCEC) Rabies Vaccine (Rabipur or equivalent) (Novartis).

INTERVENTIONS:
Biological: GSK Biological's Investigational Malaria Vaccine 257049 — All infants enrolled to group A will receive 3 doses of the experimental vaccine. The vaccine will be administered intramuscularly.
  Arms: Group A
Biological: Human Diploid Cell Vaccine (HDCV) or Purified Vero Cell Rabies Vaccine (PVRV, Verorab) (Aventis Pasteur); — To ensure consistent vaccine availability, three cell culture rabies vaccines from two manufacturers may be sourced for this trial (Aventis-Pasteur and Novartis). It will be ensured that an individual child will receive all 3 doses of cell culture rabies vaccine from the same product.
  The vaccine will be administered intramuscularly
  Arms: Group B
Biological: Purified Chick Embryo Cell Culture (PCEC) Rabies Vaccine (Rabipur or equivalent) (Novartis). — To ensure consistent vaccine availability, three cell culture rabies vaccines from two manufacturers may be sourced for this trial (Aventis-Pasteur and Novartis). It will be ensured that an individual child will receive all 3 doses of cell culture rabies vaccine from the same product.
  The vaccine will be administered intramuscularly.
  Arms: Group B

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of the candidate malaria vaccine in HIV-infected infants and children

DETAILED DESCRIPTION:
This protocol posting has been updated due to protocol Amendment 2.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* A male or female infant or child between and including 6 weeks to 17 months of age, at the time of first vaccination.
* Signed or thumb-printed informed consent obtained from the parent(s)/LAR(s) of the infant or child. Where parents/LARs are illiterate, the consent form will be countersigned by a witness.
* Subjects who the investigator believes that their parents/LARs can and will comply with the requirements of the protocol should be enrolled in the study.
* Subjects who are known to be HIV-infected (documented positive DNA PCR), whether taking HIV antiretroviral treatment (ART) or not.
* Subjects who are born following a normal gestation period.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

* Acute disease at the time of enrolment. However, the presence of an illness listed as Grade I or Grade II (WHO pediatric AIDS clinical staging) will not of itself constitute an exclusion criterion. Enrolment should be deferred if axillary temperature is >=37.5°C.
* Grade III or Grade IV abnormality on screening laboratory blood sample.
* Grade III or IV AIDS at the time of enrolment (WHO pediatric AIDS clinical staging).
* Major congenital defects.
* Planned administration/administration of a vaccine not foreseen by the study protocol prior to or within 7 days of study vaccine.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine 30 days preceding Dose°1 of study vaccine, or planned use during the study period.
* Previous participation in any other malaria vaccine trial.
* Simultaneous participation in another clinical trial including administration of experimental treatment.
* Same sex twins.
* History of allergic reactions (significant IgE-mediated events) or anaphylaxis to previous immunizations.
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.
* Child in care.

Ages: 6 Weeks to 17 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2010-07-30; Primary Completion 2013-05-24 (Actual); Study Completion 2013-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Kenya (2):
  - GSK Investigational Site, Kisian
  - GSK Investigational Site, Kisumu

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Otieno L, Oneko M, Otieno W, Abuodha J, Owino E, Odero C, Mendoza YG, Andagalu B, Awino N, Ivinson K, Heerwegh D, Otsyula N, Oziemkowska M, Usuf EA, Otieno A, Otieno K, Leboulleux D, Leach A, Oyieko J, Slutsker L, Lievens M, Cowden J, Lapierre D, Kariuki S, Ogutu B, Vekemans J, Hamel MJ. Safety and immunogenicity of RTS,S/AS01 malaria vaccine in infants and children with WHO stage 1 or 2 HIV disease: a randomised, double-blind, controlled trial. Lancet Infect Dis. 2016 Oct;16(10):1134-1144. doi: 10.1016/S1473-3099(16)30161-X. Epub 2016 Jul 7. PMID 27394191
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 112745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112745 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK257049 Group: Male and female infants and children between and including 6 weeks to 17 months of age, known to be HIV-infected, who received a 3-dose course of GSK257049 vaccine administered via intramuscular injection, for infants aged less than (<) 5 months, in the left anterolateral thigh and, for infants/children aged 5 months or more (≥ 5 months), in the left deltoid, at Days 0, 30 and 60.
- Verorab Group: Male and female infants and children between and including 6 weeks to 17 months of age, known to be HIV-infected, who received a 3-dose course of Verorab™ vaccine administered via intramuscular injection, for infants aged less than (<) 5 months, in the left anterolateral thigh and, for infants/children aged 5 months or more (≥ 5 months), in the left deltoid, at Days 0, 30 and 60.
Period: Overall Study
Arm/Group | GSK257049 Group | Verorab Group
Started | 99 | 101
Completed | 87 | 90
Not Completed | 12 | 11
Not completed — Serious Adverse Event | 5 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Migrated/moved from study area | 3 | 6
Not completed — Lost to Follow-up | 2 | 0
Not completed — Refusal | 1 | 0
Not completed — Failure to comply with study procedures | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK257049 Group | Verorab Group | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Mean (Standard Deviation); unit: Months] | 10.1 (4.99) | 9.5 (4.63) | 9.80 (4.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 45 | 102
  Male | 42 | 56 | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 99 | 101 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from 30 days before Dose 1 up to Month 14)
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 99 | 101
Participants
  Any SAE(s) | 41 | 37
  Any SAE(s) excluding Malaria | 41 | 37

2. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond (>) 20 millimeters (mm) of injection site.
Time Frame: During the 7-day post-vaccination period following each dose and across doses: Day 1 through Day 7, Month 1 through Month 1 + 7 days (Day 37), Month 2 through Month 2 + 7 days (Day 67)
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects with at least one vaccine administration documented, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 99 | 101
Participants
  Any Pain, Dose 1 | 19 | 7
  Grade 3 Pain, Dose 1 | 0 | 0
  Any Redness, Dose 1 | 6 | 3
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 11 | 4
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 95 | 100
  Any Pain, Dose 2 | 15 | 6
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 95 | 100
  Grade 3 Pain, Dose 2 | 0 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 95 | 100
  Any Redness, Dose 2 | 8 | 4
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 95 | 100
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 95 | 100
  Any Swelling, Dose 2 | 7 | 5
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 95 | 100
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 94 | 97
  Any Pain, Dose 3 | 18 | 5
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 94 | 97
  Grade 3 Pain, Dose 3 | 1 | 0
  Any Redness, Dose 3: number analyzed (Participants) | 94 | 97
  Any Redness, Dose 3 | 6 | 2
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 94 | 97
  Grade 3 Redness, Dose 3 | 0 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 94 | 97
  Any Swelling, Dose 3 | 13 | 4
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 94 | 97
  Grade 3 Swelling, Dose 3 | 1 | 0
  Any Pain, Across doses | 33 | 18
  Grade 3 Pain, Across doses | 1 | 0
  Any Redness, Across doses | 14 | 9
  Grade 3 Redness, Across doses | 0 | 0
  Any Swelling, Across doses | 26 | 13
  Grade 3 Swelling, Across doses | 1 | 0

3. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 irritability/fussiness = crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 99 | 101
Participants
  Any Drowsiness, Dose 1 | 9 | 3
  Related Drowsiness, Dose 1 | 3 | 0
  Grade 3 Drowsiness, Dose 1 | 0 | 0
  Any Irritability, Dose 1 | 21 | 12
  Related Irritability, Dose 1 | 9 | 3
  Grade 3 Irritability, Dose 1 | 0 | 0
  Any Loss of appetite, Dose 1 | 14 | 7
  Related Loss of appetite, Dose 1 | 3 | 0
  Grade 3 Loss of appetite, Dose 1 | 0 | 0
  Any Fever, Dose 1 | 31 | 20
  Related Fever, Dose 1 | 11 | 4
  Grade 3 Fever, Dose 1 | 4 | 2
  Any Drowsiness, Dose 2: number analyzed (Participants) | 95 | 100
  Any Drowsiness, Dose 2 | 10 | 6
  Related Drowsiness, Dose 2: number analyzed (Participants) | 95 | 100
  Related Drowsiness, Dose 2 | 5 | 0
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 95 | 100
  Grade 3 Drowsiness, Dose 2 | 0 | 0
  Any Irritability, Dose 2: number analyzed (Participants) | 95 | 100
  Any Irritability, Dose 2 | 22 | 12
  Related Irritability, Dose 2: number analyzed (Participants) | 95 | 100
  Related Irritability, Dose 2 | 14 | 0
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 95 | 100
  Grade 3 Irritability, Dose 2 | 0 | 0
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 95 | 100
  Any Loss of appetite, Dose 2 | 18 | 10
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 95 | 100
  Related Loss of appetite, Dose 2 | 8 | 1
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 95 | 100
  Grade 3 Loss of appetite, Dose 2 | 0 | 0
  Any Fever, Dose 2: number analyzed (Participants) | 95 | 100
  Any Fever, Dose 2 | 34 | 23
  Related Fever, Dose 2: number analyzed (Participants) | 95 | 100
  Related Fever, Dose 2 | 16 | 3
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 95 | 100
  Grade 3 Fever, Dose 2 | 2 | 0
  Any Drowsiness, Dose 3: number analyzed (Participants) | 94 | 97
  Any Drowsiness, Dose 3 | 13 | 6
  Related Drowsiness, Dose 3: number analyzed (Participants) | 94 | 97
  Related Drowsiness, Dose 3 | 6 | 2
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 94 | 97
  Grade 3 Drowsiness, Dose 3 | 0 | 0
  Any Irritability, Dose 3: number analyzed (Participants) | 94 | 97
  Any Irritability, Dose 3 | 30 | 8
  Related Irritability, Dose 3: number analyzed (Participants) | 94 | 97
  Related Irritability, Dose 3 | 19 | 2
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 94 | 97
  Grade 3 Irritability, Dose 3 | 0 | 1
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 94 | 97
  Any Loss of appetite, Dose 3 | 19 | 9
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 94 | 97
  Related Loss of appetite, Dose 3 | 8 | 1
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 94 | 97
  Grade 3 Loss of appetite, Dose 3 | 0 | 0
  Any Fever, Dose 3: number analyzed (Participants) | 94 | 97
  Any Fever, Dose 3 | 55 | 13
  Related Fever, Dose 3: number analyzed (Participants) | 94 | 97
  Related Fever, Dose 3 | 28 | 2
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 94 | 97
  Grade 3 Fever, Dose 3 | 6 | 4
  Any Drowsiness, Across doses | 22 | 15
  Related Drowsiness, Across doses | 11 | 2
  Grade 3 Drowsiness, Across doses | 0 | 0
  Any Irritability, Across doses | 46 | 25
  Related Irritability, Across doses | 29 | 5
  Grade 3 Irritability, Across doses | 0 | 1
  Any Loss of appetite, Across doses | 33 | 22
  Related Loss of appetite, Across doses | 17 | 2
  Grade 3 Loss of appetite, Across doses | 0 | 0
  Any Fever, Across doses | 74 | 46
  Related Fever, Across doses | 39 | 9
  Grade 3 Fever, Across doses | 10 | 6

4. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-day post-vaccination period (up to Day 90)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 99 | 101
Participants | 98 | 100

5. Secondary Outcome: Number of Subjects With Non-malaria Related SAEs
Description: SAEs (excluding malaria, cerebral malaria and P. falciparum parasitemia) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from 30 days before vaccine Dose 1 up to Month 14)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 99 | 101
Participants | 41 | 37

6. Secondary Outcome: Anti-circumsporozoite Protein of P. Falciparum (Anti-CS) Antibody Concentrations
Description: Anti-CS antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U/mL). The reference seropositivity cut-off value was equal to or above (≥) 0.5 EL.U/mL.
Time Frame: Prior to vaccination (PRE) and one month post Dose 3 (Month 3)
Population: The analysis was performed on the ATP population for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 81 | 73
EL.U/mL
  Anti-CS, PRE | 0.3 [0.3 to 0.4] | 0.3 [0.3 to 0.4]
  Anti-CS, Month 3: number analyzed (Participants) | 79 | 71
  Anti-CS, Month 3 | 329.2 [260.6 to 415.8] | 0.3 [0.3 to 0.3]

7. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Titers
Description: Anti-HBs antibody titers are presented as geometric mean titers (GMTs), expressed in milliinternational units per milliliter (mIU/mL).
Time Frame: Prior to vaccination (PRE) and one month post Dose 3 (Month 3)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 77 | 73
mIU/mL
  Anti-HBs, PRE | 24.1 [15.2 to 38.1] | 19.2 [12.1 to 30.6]
  Anti-HBs, Month 3: number analyzed (Participants) | 74 | 65
  Anti-HBs, Month 3 | 13637.6 [9579.7 to 19414.5] | 19.9 [12.4 to 31.9]

8. Secondary Outcome: Anti-CS Antibody Concentrations
Description: as for outcome 6
Time Frame: 12 months post Dose 3 (Month 14)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 73 | 67
EL.U/mL | 18.4 [13.3 to 25.5] | 0.3 [0.3 to 0.3]

9. Secondary Outcome: Anti-HBs Antibody Titers
Description: Anti-HBs antibody titers are presented as geometric mean titers (GMTs), expressed in mIU/mL.
Time Frame: 12 months post Dose 3 (Month 14)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 70 | 64
mIU/mL | 2294.8 [1678.2 to 3138.0] | 11.8 [7.7 to 18.1]

10. Secondary Outcome: Number of Episodes With Clinical Malaria Disease According to Primary Case Definition
Description: Primary case definition for clinical malaria: P. falciparum asexual parasitemia > 2500 parasites/μL and presence of fever (axillary temperature ≥ 37.5°C) at the time of presentation and occurring in a child who was unwell and brought for treatment to a healthcare facility.
Time Frame: From Day 0 to Month 14
Population: The analysis was performed on the ATP population for efficacy, which included all subjects included in the Total Vaccinated cohort who received all vaccinations according to protocol procedures within specified intervals that contribute time at risk in the follow-up period starting 14 days post Dose 3.
Measure: Number; unit: Episodes
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 87 | 93
Episodes | 44 | 76

11. Secondary Outcome: Number of Episodes With Severe Malaria According to Primary Case Definition
Description: The number of episodes of severe malaria of primary case definition within and outside risk period. Primary case definition for severe malaria: P. falciparum > 2500 parasites per μL and with one or more marker of disease severity and without a diagnosis of co-morbidity.
Time Frame: From Day 0 to Month 14
Population: as for outcome 10
Measure: Number; unit: Episodes
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 87 | 93
Episodes
  Episodes outside risk period | 0 | 0
  Episodes within risk period | 0 | 6

12. Secondary Outcome: Number of Subjects Affected by Prevalent Parasitemia and Prevalent Moderate Anemia
Description: The number of subjects affected by prevalent asexual P. falciparum parasitemia and prevalent moderate anemia. Moderate anemia = hemoglobin < 8 g/dL.
Time Frame: 12 months post Dose 3 (Month 14)
Population: The analysis was performed on the ATP population for efficacy, which included all subjects in the Total Vaccinated cohort who received all vaccinations according to protocol procedures within specified intervals that contribute time at risk in the follow-up period starting 14 days post Dose 3.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 87 | 93
Participants
  Prevalent parasitemia | 7 | 3
  Prevalent moderate anemia | 5 | 4

13. Secondary Outcome: Asexual P. Falciparum Parasitemia Density
Description: The number of subjects with a positive blood slide for asexual P. falciparum.
Time Frame: 12 months post Dose 3 (Month 14)
Population: The analysis was performed on children affected by prevalent parasitemia from the ATP population for efficacy, which included subjects in the Total Vaccinated cohort who received all vaccinations according to protocol procedures within specified intervals that contribute time at risk in the follow-up period starting 14 days post Dose 3.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 7 | 3
Participants | 7 | 3

14. Secondary Outcome: Prevalent Hemoglobin Level
Description: The prevalent hemoglobin level in subjects with a positive blood slide is reported as grams per deciliter (g/dl).
Time Frame: 12 months post Dose 3 (Month 14)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 87 | 93
grams per deciliter | 10.3 (1.3) | 10.1 (1.2)

15. Secondary Outcome: HIV Viral Load
Description: The HIV viral load is reported. Detectable HIV viral load: 400 or more copies/mL.
Time Frame: At baseline (PRE) and at one month (Month 3), 6 months (Month 8) and 12 months (Month 14) post Dose 3
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 99 | 101
copies/mL
  HIV viral load, PRE | 149000.00 [7490.00 to 750000.00] | 157000.00 [3630.00 to 750000.00]
  HIV viral load, Month 3 | 3125.00 [0.00 to 221500.00] | 583.50 [0.00 to 136100.00]
  HIV viral load, Month 8 | 3790.00 [0.00 to 147000.00] | 400.00 [0.00 to 103000.00]
  HIV viral load, Month 14 | 947.00 [0.00 to 99400.00] | 400.00 [0.00 to 106000.00]

16. Secondary Outcome: Percentage of CD4+ Cells
Description: The percentage of CD4+ cells is reported.
Time Frame: At baseline (PRE) and at one month (Month 3), 6 months (Month 8) and 12 months (Month 14) post Dose 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 99 | 101
Percentage
  CD4+ percentage, PRE | 27.55 (8.48) | 26.52 (8.48)
  CD4+ percentage, Month 3 | 29.70 (9.33) | 29.92 (8.67)
  CD4+ percentage, Month 8 | 32.70 (9.70) | 31.07 (9.25)
  CD4+ percentage, Month 14 | 32.80 (10.30) | 31.61 (9.56)

17. Secondary Outcome: CD4+ Absolute Cell Counts
Description: The CD4+ absolute cell counts are reported.
Time Frame: At baseline (PRE) and at 1 month (Month 3), 6 months (Month 8) and 12 months (Month 14) post Dose 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: number of cells/μL
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 99 | 101
number of cells/μL
  CD4+ absolute cell count, PRE | 2075.91 (997.81) | 2086.46 (1255.78)
  CD4+ absolute cell count, Month 3 | 2150.99 (1054.12) | 2173.04 (912.96)
  CD4+ absolute cell count, Month 8 | 2261.71 (1045.20) | 2044.51 (1014.05)
  CD4+ absolute cell count, Month 14 | 1995.36 (998.98) | 2003.70 (1027.09)

18. Secondary Outcome: World Health Organization (WHO) HIV Clinical Classification Progression
Description: Clinical staging was done at each time point according to the WHO HIV/AIDS clinical staging system. Clinical stages included:
  * "Stage 1" (asymptomatic or have persistent generalized lymphadenopathy),
  * "Stage 2" (mildly symptomatic stage - presenting with unexplained weight loss of less than 10 percent of total body weight, recurrent respiratory infections or dermatological conditions),
  * "Stage 3" (moderately symptomatic stage - presenting with weight loss of greater than 10 percent of total body weight, prolonged unexplained diarrhea or pulmonary tuberculosis, severe systemic bacterial infections or mucocutaneous conditions),
  * "Stage 4" (severely symptomatic stage which includes all of the AIDS-defining illnesses) Additional categories included "deceased" and "missing".
Time Frame: At baseline (PRE), at study months 1 (Month 1) and 2 (Month 2) and at 1 month (Month 3), 6 months (Month 8) and 12 months (Month 14) post Dose 3
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 99 | 101
Participants
  Stage 1, PRE | 81 | 82
  Stage 2, PRE | 18 | 19
  Stage 3, PRE | 0 | 0
  Stage 4, PRE | 0 | 0
  Deceased, PRE | 0 | 0
  Stage 1, Month 1 | 75 | 72
  Stage 2, Month 1 | 19 | 27
  Stage 3, Month 1 | 2 | 1
  Stage 4, Month 1 | 0 | 0
  Deceased, Month 1 | 2 | 1
  Missing, Month 1 | 1 | 0
  Stage 1, Month 2 | 79 | 77
  Stage 2, Month 2 | 15 | 20
  Stage 3, Month 2 | 1 | 2
  Stage 4, Month 2 | 0 | 0
  Deceased, Month 2 | 2 | 1
  Missing, Month 2 | 2 | 1
  Stage 1, Month 3 | 76 | 76
  Stage 2, Month 3 | 12 | 19
  Stage 3, Month 3 | 4 | 0
  Stage 4, Month 3 | 0 | 0
  Deceased, Month 3 | 2 | 2
  Missing, Month 3 | 5 | 4
  Stage 1, Month 8 | 74 | 72
  Stage 2, Month 8 | 12 | 16
  Stage 3, Month 8 | 0 | 3
  Stage 4, Month 8 | 0 | 0
  Deceased, Month 8 | 4 | 3
  Missing, Month 8 | 9 | 7
  Stage 1, Month 12 | 74 | 69
  Stage 2, Month 12 | 10 | 18
  Stage 3, Month 12 | 3 | 1
  Stage 4, Month 12 | 0 | 2
  Deceased, Month 12 | 5 | 4
  Missing, Month 12 | 7 | 7

19. Secondary Outcome: Growth Parameters: Weight, Age/Length and Middle Upper Arm Circumference for Age Z-score
Description: The following growth parameters: weight, age/length and middle upper arm circumference for age z-score are reported.
Time Frame: At baseline (PRE), at Month 3 and at study end (Month 14)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: age z-score
Arm/Group | GSK257049 Group | Verorab Group
Number analyzed (Participants) | 99 | 101
age z-score
  Height for age z-score, PRE | -1.67 (1.20) | -1.98 (1.37)
  Weight for age z-score, PRE | -1.38 (1.13) | -1.67 (1.19)
  Mid upper arm circumference z-score, PRE | -0.65 (1.13) | -0.90 (1.19)
  Height for age z-score, Month 3 | -1.91 (1.14) | -2.12 (1.16)
  Weight for age z-score, Month 3 | -1.32 (1.10) | -1.55 (1.09)
  Mid upper arm circumference z-score, Month 3 | -0.39 (1.03) | -0.65 (1.04)
  Height for age z-score, Month 14 | -1.74 (1.19) | -2.26 (1.18)
  Weight for age z-score, Month 14 | -1.10 (1.14) | -1.47 (1.02)
  Mid upper arm circumference z-score, Month 14 | -0.29 (1.13) | -0.51 (0.93)

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 30-day (Days 0-29) post vaccination period; SAEs: during the entire study period (from Day 0 up to Month 14).
Arm/Group | GSK257049 Group | Verorab Group
All-Cause Mortality (participants affected / at risk) | 5/99 | 4/101
Serious Adverse Events (participants affected / at risk) | 41/99 | 37/101
Other Adverse Events (participants affected / at risk) | 98/99 | 99/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK257049 Group (N=99) | Verorab Group (N=101)
Pneumonia (Infections and infestations) | 23 | 23
Gastroenteritis (Infections and infestations) | 21 | 19
Febrile convulsion (Nervous system disorders) | 10 | 13
Malaria (Infections and infestations) | 5 | 10
Salmonella sepsis (Infections and infestations) | 7 | 6
Malnutrition (Metabolism and nutrition disorders) | 7 | 5
Oral candidiasis (Infections and infestations) | 5 | 5
Anaemia (Blood and lymphatic system disorders) | 1 | 7
Otitis media (Infections and infestations) | 1 | 4
Pulmonary tuberculosis (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Measles (Infections and infestations) | 0 | 3
Pneumococcal sepsis (Infections and infestations) | 0 | 3
Bronchiolitis (Infections and infestations) | 0 | 2
Convulsion (Nervous system disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Helminthic infection (Infections and infestations) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tuberculosis (Infections and infestations) | 2 | 0
Abscess (Infections and infestations) | 1 | 0
Amoebiasis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Kwashiorkor (Metabolism and nutrition disorders) | 1 | 0
Meningitis haemophilus (Infections and infestations) | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4.95% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK257049 Group (N=99) | Verorab Group (N=101)
Anaemia (Blood and lymphatic system disorders) | 16 (17) | 17 (18)
Body tinea (Infections and infestations) | 6 (6) | 3 (3)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 14 (14)
Conjunctivitis (Eye disorders) | 13 (13) | 12 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 33 (51) | 23 (27)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 19 (26) | 22 (32)
Enteritis (Gastrointestinal disorders) | 26 (33) | 27 (35)
Erythema (Skin and subcutaneous tissue disorders) | 14 (20) | 9 (9)
Gastroenteritis (Infections and infestations) | 38 (58) | 41 (56)
Impetigo (Infections and infestations) | 9 (9) | 7 (7)
Irritability (Psychiatric disorders) | 46 (73) | 25 (32)
Malaria (Infections and infestations) | 22 (29) | 20 (30)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Oral candidiasis (Infections and infestations) | 11 (13) | 19 (20)
Otitis media (Infections and infestations) | 14 (14) | 15 (21)
Pain (General disorders) | 33 (52) | 18 (18)
Pneumonia (Infections and infestations) | 25 (27) | 21 (28)
Pyrexia (General disorders) | 76 (128) | 50 (67)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 9 (13)
Rash papular (Skin and subcutaneous tissue disorders) | 7 (7) | 10 (11)
Rash pruritic (Skin and subcutaneous tissue disorders) | 5 (7) | 9 (10)
Rhinitis (Infections and infestations) | 25 (27) | 18 (20)
Somnolence (Nervous system disorders) | 22 (32) | 15 (15)
Swelling (General disorders) | 26 (31) | 13 (13)
Upper respiratory tract infection (Infections and infestations) | 74 (127) | 79 (146)
Vomiting (Gastrointestinal disorders) | 5 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.